CLINICAL TRIAL: NCT06115798
Title: Laryngoscope Force During Suspension for Adenotonsillectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gianluca Bertolizio, Principle Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2023-9146
Record Dates: First submitted 2023-10-16; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Suspension laryngoscopy is a common procedure during adenoteonsillectomy (removal of adenoids and tonsils), that consists of extending the patient's neck to allow better visualization of the tonsils. Previous studies on suspension larygnoscopy have shown that the time to maximum force during this procedure predicts complications such as pain, tounge swelling and opioid requirements. Moreover, monitoring these force during laparoscopy can reduce postoperative complications. However, no study to date has investigated the force metrics during suspension laryngoscopy in the pediatric population. Therefore, in this study, the investigators aim to evaluate the relationship of force metrics during adenotonsillectomy, adenoidectomy or tonsillectomy and postoperative pain.

DETAILED DESCRIPTION:
Adenotonsillectomy is the most common surgery performed in North America (annual caseload in the United States 500,000). This procedure is performed with suspension laryngoscopy (SL), which consists in the extension of the patient's neck and concomitant lifting of the anterior oropharynx structures to allow direct visualization of the tonsils.

In adults undergoing microlaryngoscopy, the time maximum force recorded during suspension was a significant predictive variable for the development of postoperative complications such as tongue edema, pain and narcotic requirements. Force metrics during laryngoscopy vary significantly among different surgical procedures. Active intraoperative monitoring of force metrics has been shown to reduce postoperative complications in adults. Moreover, in adult cadaveric models, spinal cord compression associated with cord injury may be directly correlated with the force applied during laryngoscopy5,6. In patients with cervical instability, such as patients with Trisomy, adenotonsillectomy carries a significant risk of spinal injury, as laryngoscopy may result in C1-C2 subluxation.

To date, no data exist on force metric during suspension laryngoscopy children. The primary aim of this study is to investigate the relationship of force metrics during adenotonsillectomy, adenoidectomy or tonsillectomy and postoperative pain.

The secondary aim is to describe the force metrics in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Children ≤ 18 years old undergoing adenotonsillectomy, adenoidectomy or tonsillectomy
* Only patients whose parents are fluent in French or English will be enrolled

Exclusion Criteria:

* Any contraindication to suspension laryngoscopy
* Patient/legal guardian refusal.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Force Metrics | Measured continuously during the procedure
  Laryngoscopy suspension force
Post-operative negative behaviors (pain, emergence delirium and hypoactive delirium) | 1 hour after the produce
  Laryngoscopy suspension force as a tool to predict post-operative negative behaviors

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Bertolizio, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada